CLINICAL TRIAL: NCT03235557
Title: Robotic Radiation Treatment of Prostate Cancer Patients Aged 70 y or More
Brief Title: CyberKnife for Prostate Cancer Patients Aged 70 y or More
Acronym: ProRobot
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse, Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: CYM Prostate CFB 1
Record Dates: First submitted 2015-01-15; First posted 2017-08-01 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; radiation; stereotactic; CyberKnife; elderly
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Robotic Stereotactic Radiation treatment of prostatic adenocarcinoma of the elderly.

Inclusion criteria : T1-T3b, MRI pelvic nodes negative, M0, any Gleason Score, PSA (Prostate Specific Antigen) <30ng/ml.

Dose : 36.25 Gy in 5 fractions, in 10 days, considering CAPRA Scores≤5 AND 37.5 Gy in 5 fractions, in 10 days, considering CAPRA Scores>5.

Primary objective : acute and late toxicity evaluation at 36 months. Secondary objectives : PSA and MRI response.

DETAILED DESCRIPTION:
Robotic Stereotactic Radiation treatment of prostatic adenocarcinoma of the elderly.

Rationale : Half of the prostatic adenocarcinoma are diagnosed in the elderly but until now curative treatments were not proven to increase overall survival rates. Therefore, very short, comfortable and safe treatments have to be designed to increase the pelvic control of the disease. Moreover, the alpha/beta ratio of the disease ≤3Gray is in favour of using hypofractionation schemes.

Primary objective : acute and late toxicity evaluation at 36 months. Secondary objectives : PSA and MRI response and quality of life evaluation.

Inclusion criteria : T1-T3b, MRI pelvic nodes negative, M0, any Gleason Score, PSA<30ng/ml.

Dose : 36.25 Gray in 5 fractions, in 10 days, considering CAPRA Score≤5 AND 37.5 Gray in 5 fractions, in 10 days, considering CAPRA Scores>5.

Doses to the Organs At Risk (OAR) : Rectum wall : V36.25<2%, V27<20%, V23<30%, V20<35%. Bladder wall : V36.25<2%, V27<20%, V20<35%. Considering specifically the prescription of 37.5 Gray, the rectum and bladder wall: V37.5<2%. Anytime, hot spots of 105 % of the prescription dose must avoid the urethra.

Evaluation criteria : CTCAEV4 (Common Toxicity Criteria for Adverse Events, version4), PSA, multiparametric MRI, IPSS (International Prostate Score Symptom) and IIEF5 (International Index of Erectile Function).

Methodolgy : this is a three step prospective, observational study of 20 patients each step. Before moving to the next step, the severe acute or late toxicity at a median follow-up of 1 year must remain below 5% each.

ELIGIBILITY:
Inclusion Criteria:

* T1-T3b,
* MRI pelvic nodes negative,
* M0,
* any Gleason Score,
* PSA<30ng/ml,
* WHO (World Health Organisation) score<2, IPSS≤15,
* maximal urinary flow rate ≥15ml/s,
* mean urinary flow rate ≥5ml/s,
* multiparametric prostatic and pelvis MRI

Exclusion Criteria:

* Prostatic volume > 100cc,
* TURP (transurethral prostatectomy) <3 y,
* any recurrent prostatitis within the last 3 years,
* collagenose diseases,
* ulcero-haemorrhagic rectocolitis or
* crohn diseases

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients suffering prostatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Acute and late toxicity (Using the CTCAEv4) | During 36 months after treatment
  Using the CTCAEv4

SECONDARY OUTCOMES:
PSA evaluation | at 4 and 6 months, than every 6 months for 3 years
  PSA Dosage
Digital rectal exam | at 6, 12, 24 and 36 months
  Clinical examination (digital rectal exam)
Birads score evaluation | at 36 months
  Multiparametric prostatic MRI
IPSS evaluation | at 12, 24 and 36 months
  IPSS score
IIEF5 evaluation | at 12, 24 and 36 months
  IIEF5 score

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nickers, MD, PhD, Study Chair — Centre Francois Baclesse; Michel Untereiner, MD, Study Director — Centre Francois Baclesse
Locations (1):
- Centre Francois Baclesse, Esch-sur-Alzette, Luxembourg

REFERENCES:
- [Result] Nickers P, Hermesse J, Deneufbourg JM, Vanbelle S, Lartigau E. Which alpha/beta ratio and half-time of repair are useful for predicting outcomes in prostate cancer? Radiother Oncol. 2010 Dec;97(3):462-6. doi: 10.1016/j.radonc.2010.06.006. Epub 2010 Aug 17. PMID 20724012
- [Result] Boike TP, Lotan Y, Cho LC, Brindle J, DeRose P, Xie XJ, Yan J, Foster R, Pistenmaa D, Perkins A, Cooley S, Timmerman R. Phase I dose-escalation study of stereotactic body radiation therapy for low- and intermediate-risk prostate cancer. J Clin Oncol. 2011 May 20;29(15):2020-6. doi: 10.1200/JCO.2010.31.4377. Epub 2011 Apr 4. PMID 21464418
- [Result] King CR, Brooks JD, Gill H, Presti JC Jr. Long-term outcomes from a prospective trial of stereotactic body radiotherapy for low-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):877-82. doi: 10.1016/j.ijrobp.2010.11.054. Epub 2011 Feb 6. PMID 21300474